CLINICAL TRIAL: NCT04511156
Title: A Training Package for the World Health Organization Foundational Helping Skills in Mental Health and Psychosocial Support Services: Study Protocol for A Mixed-Methods Evaluation
Brief Title: Ensuring Quality in Psychological Support-Foundational Helping Skills
Acronym: EQUIP-FHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: World Health Organization (Other); Transcultural Psychosocial Organization Nepal (Other); Socios En Salud Sucursal, Peru (Other); HealthRight International (Unknown)
Responsible Party: Principal Investigator, Brandon A Kohrt, MD, PhD, Associate Professor, George Washington University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EQUIP-FHS
Record Dates: First submitted 2020-07-29; First posted 2020-08-13 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Psychological Distress
Keywords: Competency; Training; Communication skills; Empathy

STUDY DESIGN:
Intervention Model Description: This study is a single group, multi-site, uncontrolled before- and-after trial, which will evaluate the effectiveness of a training intervention to improve foundational helping skills in non-specialists naïve to mental health and psychosocial support. We will compare change in trainees' foundational helping skills competency scores from pre-training (baseline) to post-training, as well as knowledge, attitude, and self-efficacy scores. We will also explore the feasibility, acceptability, and perceived benefit of the Foundational Helping Skills training package for remote and in-person delivery. The study will be conducted in three country settings, Nepal, Perú and Uganda. The study design will be the same in all three country sites.
Masking Description: Raters of competency will watch video-taped role plays and they will be blinded as to whether the role plays were conducted pre- or post-training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Foundational Helping Skills (Experimental): The Foundational Helping Skills training will be intervention to be evaluated in this study. The Foundational Helping Skills is a flexible curriculum, with an approximate 3-day (20 hour) duration to be modified based on context and personnel. The Foundational Helping Skills is a human-centered design competency-based training in foundational helping skills. The training curriculum has been developed in a modular format, with each module relating to specific foundational helping skills (e.g., non-verbal communication, confidentiality, etc). The training curriculum can be found. The general training outline includes two days of foundational helping skill modules, brief role-play competency assessments at the end of each foundational helping skills training day to inform trainers which competencies need remediation, and a half-day of training that involves a remediation of the specific foundational helping skills that have been identified via the brief role-play assessments.
  Interventions: Other: Foundational Helping Skills

INTERVENTIONS:
Other: Foundational Helping Skills — Each site will implement three waves of Foundational Helping Skills training. Each training will include 12 trainees each, with a minimum of 2 trainers per training. Each site will include pre and post research days, where they will collect primary and secondary outcomes with support from research staff (trained raters, actors, and qualitative researcher). Each site will qualitatively assess the training after the first wave to identify any areas for modification, and after the second and third waves to develop recommendations for future implementation.

SUMMARY:
There is lack of feasible and effective curricula that can rapidly be taught on basic mental health and psychosocial helping skills. Through the World Health Organization Ensuring Quality in Psychological Support initiative, a curriculum has been developed focusing on common factors in mental health and psychosocial support, such as verbal and nonverbal communication skills, empathy, rapport building, and promoting hope and expectancy of change. To minimize training burden and maximize effectiveness, this has been designed as a competency-based training wherein target competencies are evaluated throughout the training so that it can tailored to trainees preexisting skills, rather than using a one-size-fits-all approach to the training. The training duration and content is modular and flexible, with approximately 16 hours of modules content. The investigator's goal is to conduct a mixed-methods evaluation of the foundational helping skills program. In three countries, Nepal, Peru, and Uganda, two trainers (total n=6 across countries) and 36 service providers (total n=108 across countries) without prior training in mental health and psychosocial support skills will receive the training. Their competency in foundational helping skills will be evaluated prior to training using an objective structured clinical examination approach with standardized role plays using trained raters and actor (i.e., standardized clients). Role play ratings will be made using the ENhancing Assessment of Common Therapeutic factors. In addition, trainees knowledge and perceived self-efficacy in foundational helping skills will be evaluated pre- and post-training. Trainers and trainees will also participate in qualitative interviews regarding feasibility, acceptability, and perceived benefit of the foundational helping skills program. A mixed methods evaluation of the foundational helping skills curriculum will help to inform further revision of the materials on the Ensuring Quality in Psychological Support platform. Determination of the change in skills, knowledge, and self-efficacy will identify effective components of the platform and areas for further refinement. Ultimately, an effective training program in foundational helping skills will contribute to improved health, psychological, and social services around the world.

DETAILED DESCRIPTION:
The World Health Organization Ensuring Quality in Psychological Support program is currently developing a Universal Foundational Helping Skills Training package. This training package will be freely available for use by all health professionals and other service providers seeking to develop basic skills in mental health and psychosocial support. These foundational helping skills are based upon common factors in the mental health and psychological services, which have been widely researched and identified as essential and universal prerequisites for the effective delivery of any psychosocial or psychological components in health interventions. These are also foundational skills are also part of the competencies for non-specialists to deliver psychological interventions in global mental health. Competent use of these skills by providers improves outcomes for people accessing all fields of health services--ranging from surgery to pain clinics--support greater treatment adherence. A foundational helping skills training curriculum is needed to promote competency in the provision of warm and trusting relationships between health care providers and people accessing health services. Other foundational helping skills include rapport building, the demonstration of empathy, using culturally or age-appropriate terminology and concepts for distress, and ensuring communication of hope. This training guidance will fill the gap many training programs for providers who are not mental health specialists, and the training guidance will be feasible for implementation in low-resource settings. The training will be aligned with the World Health Organization competency framework for the health sector that is under development, which stipulates foundational helping skills as essential for all health cadres. The World Health Organization Universal Foundational Helping Skills Training package has the potential to improve competency for basic mental health and psychosocial support services delivered by any health cadres. This training package, alongside other quality improvement activities, will lead to more effective delivery of quality care for clients and will be one step closer to achieving the global communities' and World Health Organization's goal of universal health care. The goal of this study is to conduct a mixed-methods evaluation of the Foundational Helping Skills curriculum by observing outcomes for trainees in the program who not have prior mental health and psychosocial support skills training.

ELIGIBILITY:
Inclusion Criteria:

* All trainees participating in the training must be over 18 years old,
* have no prior experience in mental health and psychosocial support care or delivery.
* Trainees need to have fluency in the language in which the trainings will be conducted: Nepali in Nepal, Spanish in Peru, and English in Uganda.
* In sites where the training will be delivered remotely, access to online service and device with video and audio capabilities will be expected.

Exclusion Criteria:

* Trainees will not be able to participate in the training if they are under 18 years old,
* have experience in mental health and psychosocial support care of delivery or
* have completed education in a mental health related field or similar training or delivery (e.g., completed psychology degree).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Enhancing Assessment of Common Therapeutic Factors; Unabbreviated scale title: "Enhancing Assessment of Common Therapeutic Factors" | immediately after the foundational helping skills training
  15-item objective structured clinical examination using a role play, minimum value = 15, maximum value = 60, higher score means greater competency

SECONDARY OUTCOMES:
Foundation Helping Skills Knowledge Test; Unabbreviated scale title: "Foundation Helping Skills Knowledge Test" | immediately after the foundational helping skills training
  Multiple choice test for each of the common factors competencies; minimum value=0, maximum value = 30, scores are reported of percentages of total, minimum = 0%, maximum = 100%, higher scores mean more knowledge of foundational helping skills
Counselor Activity Self-Efficacy Scales; Unabbreviated scale title: "Counselor Activity Self-Efficacy Scales" | immediately after the foundational helping skills training
  15-item self-efficacy scale for counseling skills; minimum value = 0, maximum value = 135, higher scores mean more perceived self-efficacy in counselor skills

CONTACTS AND LOCATIONS:
Overall Officials: Alison Schafer, PhD, Principal Investigator — World Health Organization
Locations (3):
- Transcultural Psychosocial Organization Nepal, Kathmandu, Nepal
- Socios en Salud Sucursal Peru, Lince, Peru
- HealthRight International Uganda, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared after publication of primary results.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Materials will be shared after publication of primary results.
Access Criteria: Contact investigators.